CLINICAL TRIAL: NCT06101927
Title: SPECT Imaging of Prostate-Specific Membrane Antigen Using Labeled Technetium-99m BQ0413 ([99mTc]Tc- BQ0413) in Prostate Cancer Patients
Brief Title: Molecular Imaging of Prostate-Specific Membrane Antigen Using Labeled Technetium-99m BQ0413
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: [99mTc]Tc- BQ0413
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
Keywords: Prostate-Specific Membrane Antigen; Prostate cancer; [99mTc]Tc-BQ0413; SPECT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Prostate cancer 50 mkg (Experimental): At least five (5) evaluable subjects with prostate cancer with [99mTc]Tc-BQ0413 (50 mkg)
  Interventions: Drug: Whole body study and SPECT with [99mTc]Tc-BQ0413
- Experimental: Prostate cancer 100 mkg (Experimental): At leaAt least five (5) evaluable subjects with prostate cancer with [99mTc]Tc-BQ0413 (100 mkg)
  Interventions: Drug: Whole body study and SPECT with [99mTc]Tc-BQ0413

INTERVENTIONS:
Drug: Whole body study and SPECT with [99mTc]Tc-BQ0413 — One single intravenous injection of [99mTc]Tc-BQ0413, followed by gamma camera imaging after 2, 4, 6 and 24 hours.
  Other Names: Diagnostic Test:

SUMMARY:
The study should evaluate the biological distribution of [99mTc]Tc-BQ0413 in patients with prostate cancer.

The primary objective are:

1. To assess the distribution of [99mTc]Tc- BQ0413 in normal tissues and tumors at different time intervals.
2. To evaluate dosimetry of [99mTc]Tc- BQ0413.
3. To study the safety and tolerability of the drug [99mTc]Tc- BQ0413 after a single injection in a diagnostic dosage.

The secondary objective are:

1. To compare the obtained [99mTc]Tc- BQ0413 SPECT imaging results with the data of CT and/or MRI and/or ultrasound examination and immunohistochemical (IHC) studies in prostate cancer patients.

DETAILED DESCRIPTION:
The overall goal is to study the effectiveness of SPECT imaging prostate cancer patients Using technetium-99m labeled BQ0413.

Phase I of the study:

Biodistribution of [99mTc]Tc-BQ0413 in patients with prostate cancer.

The main objectives of the study:

1. To evaluate the distribution of [99mTc]Tc-BQ0413 in normal tissues and tumors in patients with prostate cancer at different time intervals.
2. To evaluate dosimetry of [99mTc]Tc-BQ0413 based on the pharmacokinetic parameters of the drug after a single intravenous administration.
3. To study the safety of use and tolerability of the drug [99mTc]Tc-BQ0413 after a single intravenous administration in a diagnostic dosage.

Additional research tasks:

1. To conduct a comparative analysis of the diagnostic information obtained in the visualization of prostate cancer by SPECT using [99mTc]Tc-BQ0413 with data obtained by CT and/or MRI and/or ultrasound examination and immunohistochemical (IHC) research of postoperative material.

Methodology:

Open-label, exploratory, single centre study. The subjects will receive a single injection of the labeled tracer.

ELIGIBILITY:
Inclusion Criteria:

* Subject is > 18 years of age
* Clinical and radiological diagnosis of prostate cancer with histological verification.
* White blood cell count: > 2.0 x 10^9/L
* Haemoglobin: > 80 g/L
* Platelets: > 50.0 x 10^9/L
* Bilirubin =< 2.0 times Upper Limit of Normal
* Serum creatinine: Within Normal Limits
* Blood glucose level not more than 5.9 mmol/L
* Subject is capable to undergo the diagnostic investigations to be performed in the study
* Informed consent

Exclusion Criteria:

* Active current autoimmune disease or history of autoimmune disease
* Active infection or history of severe infection within the previous 3 months (if clinically relevant at screening)
* Known HIV positive or chronically active hepatitis B or C
* Administration of other investigational medicinal product within 30 days of screening
* Ongoing toxicity > grade 2 from previous standard or investigational therapies, according to US National Cancer Institute's

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men
Enrollment: 10 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Gamma camera-based whole-body [99mTc]Tc-BQ0413 uptake value (%) | 24 hours
  Whole-body [99mTc]Tc-BQ0413 uptake coinciding with normal organs and tissues will be assessed using gamma camera and calculated as percentage (%) of the injected dose of the radiopharmaceutical
SPECT-based [99mTc]Tc-BQ0413 value in tumor lesions (counts) | 6 hours
  [99mTc]Tc-BQ0413 uptake coinciding with tumor lesions will be assessed using single-photon emission computed tomography and measured in counts
SPECT-based [99mTc]Tc-BQ0413 uptake value (counts) | 6 hours
  Focal uptake of [99mTc]Tc-BQ0413 in the regions without pathological findings will be assessed with SPECT and measured in counts
Tumor-to-background ratio (SPECT) | 6 hours
  The SPECT-based tumor-to-background ratio will be calculated as follows: the value of [99mTc]Tc-BQ0413 uptake coinciding with tumor lesions (counts) will be divided by the value of [99mTc]Tc-BQ0413 uptake coinciding with the regions without pathological findings (counts)

SECONDARY OUTCOMES:
Percent of cases with abnormal findings relative to baseline [Safety and Tolerability] | 24 hours
  The safety attributable to [99mTc]Tc-BQ0413 injections will be evaluated based on the assessments of physical examination, vital signs, and ECG (percent of cases with abnormal findings relative to baseline)
Percent of participants with abnormal laboratory values that are related to diagnostic imaging procedure [Safety and Tolerability] | 24 hours
  The safety attributable to [99mTc]Tc-BQ0413 injections will be evaluated based on the blood and urine laboratory tests (percent of cases with abnormal findings relative to baseline)
Percent of participants with adverse events that are related to diagnostic imaging procedure [Safety and Tolerability] | 24 hours
  The safety attributable to [99mTc]Tc-BQ0413 injections will be evaluated based on the rate of adverse events (percent)
Percent of participants requiring administration of medication due to side effects that are related to diagnostic imaging procedure [Safety and Tolerability] | 24 hours
  The safety attributable to [99mTc]Tc-BQ0413 injections will be evaluated based on the rate of administration of concomitant medication (percent)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir I Chernov, MD,Prof, Study Director — Tomsk NRMC
Locations (1):
- TomskNRMC, Tomsk, Russia